CLINICAL TRIAL: NCT02341612
Title: Effects of Different Cold Therapy Modalities on Muscular Recovery and Inflammatory Responses Following Exercise-induced Muscle Damage in Healthy Men
Brief Title: Cold Therapy in the Treatment of Exercise-induced Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Angelina Freitas Siqueira, Angelina Freitas Siqueira, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP/FS-UnB 234/13
Record Dates: First submitted 2014-12-16; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Cryotherapy Effect
Keywords: exercise-induced muscle damage; skeletal muscle injury recovery; cryotherapy; recovery of function; rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- single exposure at 5°C in CWI (Experimental): The subjects of this group performed cold water immersion (CWI) immediately after exercise-induced muscle damage (EIMD) a single exposure at 5°C for 20 minutes.
  Interventions: Other: single exposure at 5°C in CWI
- single exposure at 15°C in CWI (Experimental): The subjects of this group performed CWI immediately after EIMD a single exposure at 15°C for 20 minutes.
  Interventions: Other: single exposure at 15°C in CWI
- multiple exposures at 10°C in CWI (Experimental): The subjects of this group performed CWI immediately, 24h, 48h and 72h after EIMD (once a day) for 20 minutes.
  Interventions: Other: multiple exposures at 10°C in CWI
- whole body criotherapy (WBC) (Experimental): The whole body criotherapy (WBC) group remained in the cabin immediately after EIMD for 3 minutes.
  Interventions: Other: whole body cryotherapy (WBC)
- passive recovery (Experimental): The control group was not exposed to treatment after the EIMD protocol.
  Interventions: Other: passive recovery

INTERVENTIONS:
Other: single exposure at 5°C in CWI — The subjects of this group performed cold water immersion immediately after exercise-induced muscle damage (EIMD) a single exposure at 5°C for 20 minutes.
  Arms: single exposure at 5°C in CWI
Other: single exposure at 15°C in CWI — The subjects of this group performed CWI immediately after EIMD a single exposure at 15°C for 20 minutes.
  Arms: single exposure at 15°C in CWI
Other: multiple exposures at 10°C in CWI — The subjects of this group performed CWI immediately, 24h, 48h and 72h after EIMD (once a day) for 20 minutes.
  Arms: multiple exposures at 10°C in CWI
Other: whole body cryotherapy (WBC) — The whole body criotherapy (WBC) group remained in the cabin immediately after EIMD for 3 minutes.
  Arms: whole body criotherapy (WBC)
Other: passive recovery — The control group was exposed to treatment after the EIMD protocol.
  Arms: passive recovery

SUMMARY:
Subjects were randomly placed in five groups: (1) single exposure at 5°C in cold water immersion, (2) single exposure at 15°C in cold water immersion, (3) multiple exposures at 10°C in cold water immersion, (4) whole body cryotherapy (WBC) at 110°C and (5) passive recovery (control group). The single exposure groups performed cold water immersion immediately after exercise-induced muscle damage (EIMD) for 20 minutes. The multiple exposures group performed cold water immersion immediately, 24h, 48h and 72h after EIMD (once a day) for 20 minutes. The WBC group remained in the cabin immediately after EIMD for 3 min. The control group was not exposed to treatment after the EIMD protocol. The subjects were asked to visit the laboratory on seven occasions. The first visit was the familiarization of the subjects with experimental procedures and their anthropometric assessment. One week after familiarization, on visit two, volunteers performed the exercise-induced muscle damage (EIMD) protocol and they were allocated to one of experimental groups. Indirect markers of muscle damage and inflammatory responses were evaluated at baseline (pre), immediately post, 24h, 48h, 72h, 96h, and 168h following the EIMD protocol by measuring anterior thigh muscle swelling, isometric knee extensors peak torque, knee extensors muscle soreness, countermovement vertical jump and blood sample analyzes.

DETAILED DESCRIPTION:
To avoid circadian influences, subjects were asked to visit the laboratory always at the same time of day. Volunteers were asked to not perform any vigorous physical activities or unaccustomed exercise during the experiment period. In addition, they were instructed not to intake medications or supplements during the study.

ELIGIBILITY:
Inclusion Criteria:

* College students were eligible for inclusion.

Exclusion Criteria:

* Exclusion criteria included a history of eccentric quadriceps exercise in the past 3 months
* A history of quadriceps muscle tear
* Neurological disease involving the lower limbs
* Current lower-limb musculoskeletal injury and thigh skinfold thickness >20 mm..
* Participants with potential vascular problems which cold therapy is contraindicated (eg, diagnoses of diabetes or Raynaud's disease) were also excluded

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change of knee extensors muscle maximal isometric voluntary contraction during 168h post exercise-induced muscle damage (EIMD), assessed using isokinetic dynamometer | at baseline (pre) and at 0, 24, 48, 72, 96, and 168 hours after exercise-induced muscle damage.

SECONDARY OUTCOMES:
Change of the anterior thigh muscle swelling during 168h post EIMD, assessed using ultrasound device | at baseline (pre) and at 0, 24, 48, 72, 96, and 168 hours after exercise-induced muscle damage.
Change of the knee extensors muscle soreness during 168h post EIMD, assessed using a Visual Analogue Scale | at baseline (pre) and at 0, 24, 48, 72, 96, and 168 hours after exercise-induced muscle damage.
Change of inflammatory response (Tumor Necrosis Factor-α, interleukin-6, interleukin-10, interleukin-1β, interleukin-1ra) during 168h post EIMD, assessed by blood sample analyzes | at baseline (pre) and at 0, 24, 48, 72, 96, and 168 hours after exercise-induced muscle damage.
Change on the performance of countermovement vertical jump during 168h post EIMD, assessed using a force plate | at baseline (pre) and at 0, 24, 48, 72, 96, and 168 hours after exercise-induced muscle damage.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Brasília, Brasília, Federal District, Brazil